CLINICAL TRIAL: NCT02836418
Title: An Open-Label Extension Study to Evaluate the Long-Term Safety, Tolerability, and Biological Activity of ATYR1940 in Patients With Limb Girdle and Facioscapulohumeral Muscular Dystrophy
Brief Title: Study to Evaluate the Long-Term Safety, Tolerability, and Biological Activity of ATYR1940 in Participants With Limb Girdle and Facioscapulohumeral Muscular Dystrophy (FSHD)
Acronym: FSHD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: aTyr Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATYR1940-C-006
Record Dates: First submitted 2016-06-30; First posted 2016-07-19 (Estimated); Results first posted 2023-12-22 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Facioscapulohumeral Muscular Dystrophy; Limb Girdle Muscular Dystrophy
Keywords: FSHD; LGMD
MeSH Terms: conditions — Muscular Dystrophy, Facioscapulohumeral; Muscular Dystrophies, Limb-Girdle

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ATYR1940 (Experimental): Participants will receive ATYR1940 up to 3.0 milligrams per kilograms (mg/kg) intravenous (IV) infusion once weekly until approval of ATYR1940, discontinuation of its development, the study was closed by the Sponsor, or a criterion for study drug discontinuation (up to 34 weeks).
  Interventions: Drug: ATYR1940

INTERVENTIONS:
Drug: ATYR1940 — Concentrate for solution for infusion

SUMMARY:
ATYR1940-C-006 is a multi-national, multicenter study being conducted at centers in the United States (US) and Europe who participated in Study ATYR1940-C-003 (Stage 1 only) or Study ATYR1940-C-004 (that is, the parent studies).

DETAILED DESCRIPTION:
Study ATYR1940-C-006 is a multi-national, multi-center, open-label extension study designed to evaluate the long-term safety, effects on muscle, and pharmacodynamics of ATYR1940 in participants with Limb-girdle muscular dystrophy (LGMD) or FSHD previously treated in the Study ATYR1940-C-003 (Stage 1 only) or Study ATYR1940-C-004 that is, the parent studies). This study will be conducted at the same study centers at which participants were enrolled in the parent studies.

Participants who completed the treatment period in the parent study and, in the Investigator's opinion, demonstrated acceptable tolerability of ATYR1940, are considered by the Investigator to be compliant with ATYR1940 and the study procedures, and do not meet any criterion for ATYR1940 discontinuation are eligible for participation in the current study, contingent upon Investigator and participant agreement to continue ATYR1940 treatment.

For the first 12 weeks in this extension study, participants will receive ATYR1940 at the highest tolerated dose received in the parent study; no dose adjustments are allowed during this 12-week period. After 12 weeks, if the participant is demonstrating good tolerability, the ATYR1940 dose may be increased on a participant-specific basis at the Investigator's discretion, in consultation with the Sponsor and Medical Monitor. ATYR1940 dose increases to >3.0 mg/kg are not permissible.

All participants will receive ATYR1940 on a weekly basis in this study, regardless of the frequency of dosing in the parent study. ATYR1940 will be administered via intravenous (IV) infusion over 90 minutes. If medically indicated, the infusion duration and volume may be adjusted at the Investigator's discretion in consultation with the Medical Monitor and Sponsor.

ELIGIBILITY:
Inclusion Criteria:

1. Enrolled in and completed the treatment period in the parent study.
2. Demonstrated, in the Sponsor's and Investigator's opinions, acceptable tolerability of ATYR1940.
3. In the Investigator's opinion, participant has shown acceptable compliance with ATYR1940 and the study procedures in the parent study and is willing and able to comply with all procedures in the current study.
4. Is, in the opinion of the Investigator and Sponsor, a suitable candidate for continued ATYR1940 treatment.
5. Provide written informed consent or assent after the nature of the study has been explained and prior to the performance of any research-related procedures.

Exclusion Criteria:

1. Is expected to require treatment with curcumin or systemic albuterol (intermittent inhaled albuterol is permissible) during study participation; or use of a product that putatively enhances muscle growth (for example, insulin-like growth factor, growth hormone) or activity (for example, Coenzyme Q, Coenzyme A, creatine, L-carnitine) on a chronic basis; or statin treatment initiation or significant adjustment to statin regimen (stable, chronic statin use is permissible).
2. Planned to receive any vaccination during study participation.
3. Abnormal baseline findings, medical condition(s), or laboratory findings that, in the Investigator's opinion, might jeopardize the participant's safety or decrease the chance of obtaining satisfactory data needed to achieve the objectives of the study.
4. Evidence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematological, metabolic, dermatological, or gastrointestinal disease, or has a condition that requires immediate surgical intervention, other treatment, or may not allow safe participation.
5. If female and of childbearing potential (premenopausal and not surgically sterile), has a positive pregnancy test at entry or is unwilling to use contraception from the time of entry through the 3-month Follow-up visit. Acceptable methods of birth control include abstinence, barrier methods, hormones, or intra-uterine device.
6. If male, is unwilling to use a condom plus spermicide during sexual intercourse from the time of entry through the 1 month Follow-up visit.

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2016-07-13 (Actual); Primary Completion 2017-04-18 (Actual); Study Completion 2017-04-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (3):
  - University of California, Irvine, ALS and Neuromuscular Center, Irvine, California
  - Stanford University, Stanford, California
  - University of Utah, Salt Lake City, Utah
- Rigshospitalet, University of Copenhagen, Copenhagen, Denmark
- Foundation IRCCS Neurological Institute Carlo, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who participated in and completed the treatment period and were considered to be compliant with the study drug by the Investigator in the parent studies (ATYR1940-C-003 [NCT02603562] or ATYR1940-C-004 [NCT02579239]) were eligible for participation in this study. Note that only data for this study are reported in this Results Record. Data for the parent studies (ATYR1940-C-003 [NCT02603562] and ATYR1940-C-004 [NCT02579239]) are reported in the respective Results Records.
Pre-assignment Details: When a participant transferred from the parent study to this extension study, the duration between the last ATYR1940 dose in the parent study and first ATYR1940 dose in this extension study was to be 1 week; however, a maximum duration of 3 weeks was permissible.
Groups:
- ATYR1940: Participants received ATYR1940 up to 3.0 milligrams per kilograms (mg/kg) intravenous (IV) infusion once weekly until approval of ATYR1940, discontinuation of its development, the study was closed by the Sponsor, or a criterion for study drug discontinuation was met (up to a maximum of 34 weeks).
Period: Overall Study
Arm/Group | ATYR1940
Started | 8
Received at Least One Dose of Study Drug | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Cumulative Safety population included all participants who received at least 1 full or partial dose of ATYR1940 in the current study (Study ATYR1940-C-006) and had a post-infusion safety observation since enrollment in parent studies, but with cumulative data from both the parent studies and the current study.
Groups:
- ATYR1940: Participants received ATYR1940 up to 3.0 mg/kg IV infusion once weekly until approval of ATYR1940, discontinuation of its development, the study was closed by the Sponsor, or a criterion for study drug discontinuation was met (up to a maximum of 34 weeks).
Arm/Group | ATYR1940
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.0 (15.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: TEAEs were defined as adverse events (AEs) with an onset following administration of the first dose of study drug. AEs were defined as any untoward medical occurrence in a participant administered study drug and that does not necessarily have a causal relationship with the study drug. Worsening of a pre-existing medical condition should have been considered an AE if there was either an increase in severity, frequency, or duration of the condition or an association with significantly worse outcomes. SAEs were defined as any AE that, in the view of either the Investigator or Sponsor, resulted in any of the following outcomes as fatal, life-threatening, required in-participant hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, a congenital anomaly/birth defect, an important medical event. A summary of all SAEs and Other AEs (nonserious) regardless of causality is located in 'Reported Adverse Events' Section.
Time Frame: Up to End of Study (up to approximately Week 39)
Population: Safety population was defined as all participants who received at least 1 full or partial dose of ATYR1940 in the current study (Study ATYR1940-C-006) and had a post-infusion safety observation since enrollment in parent studies.
Measure: Count of Participants; unit: Participants
Arm/Group | ATYR1940
Number analyzed (Participants) | 8
Participants
  TEAEs | 7
  SAEs | 0

2. Primary Outcome: Number of Participants With Positive Anti-Drug Antibodies (ADA)
Description: Summarized titers are reported below.
Time Frame: Up to End of Study (up to approximately Week 39)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | ATYR1940
Number analyzed (Participants) | 8
Participants | 3

3. Primary Outcome: Number of Participants With a Jo-1 Antibody (Ab) Test Result ≥1.5 Units/Milliliter (U/mL)
Description: Participants with Jo-1 Ab levels ≥1.5 U/mL were to be discontinued from dosing of the study drug.
Time Frame: Up to End of Study (up to approximately Week 39)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | ATYR1940
Number analyzed (Participants) | 8
Participants | 2

4. Primary Outcome: Number of Participants With a Clinical Laboratory Abnormality Leading to an AE
Description: Laboratory parameters included hematology (hematocrit, hemoglobin, red blood cell count, white blood cell count neutrophils, lymphocytes, monocytes, eosinophils, basophils, and platelet count); serum chemistries (blood urea nitrogen, creatinine, total bilirubin, aspartate aminotransferase, alanine aminotransferase, gamma-glutamyl transferase, alkaline phosphatase, total protein, sodium, potassium, bicarbonate, calcium, chloride, magnesium, inorganic phosphate, creatine kinase, lactate dehydrogenase, C-reactive protein, troponin, myoglobin, insulin-like growth factor 1, and cholesterol [nonfasting]); and urinalysis (color, pH, specific gravity, protein, glucose, ketones, and blood). Clinically significant laboratory abnormalities were based upon Investigator's discretion. A summary of all Serious Adverse Events and Other Adverse Events (nonserious) regardless of causality is located in the 'Reported Adverse Events' Section.
Time Frame: Up to End of Study (up to approximately Week 39)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | ATYR1940
Number analyzed (Participants) | 8
Participants | 1

5. Primary Outcome: Number of Participants With a Clinically Significant Pulmonary Function Event Resulting in a TEAE
Description: Pulmonary evaluations included pulmonary function tests and pulse oximetry. Clinically significant changes were to be reported as adverse events. A summary of all Serious Adverse Events and Other Adverse Events (nonserious) regardless of causality is located in the 'Reported Adverse Events' Section.
Time Frame: Up to End of Study (up to approximately Week 39)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | ATYR1940
Number analyzed (Participants) | 8
Participants | 0

6. Primary Outcome: Number of Participants With a Clinically Significant Electrocardiogram (ECG) Abnormality Leading to a TEAE
Description: ECG parameters that were evaluated included heart rate and PR, QR, and QT intervals. A clinically significant ECG abnormality was based upon the Investigator's discretion. A summary of all Serious Adverse Events and Other Adverse Events (nonserious) regardless of causality is located in the 'Reported Adverse Events' Section.
Time Frame: Up to End of Study (up to approximately Week 39)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | ATYR1940
Number analyzed (Participants) | 8
Participants | 2

7. Primary Outcome: Number of Participants With Vital Sign Abnormality Resulting in a TEAE
Description: The vital sign parameters that were evaluated included heart rate, systolic and diastolic blood pressure, and respiration rate as well as temperature. A summary of all Serious Adverse Events and Other Adverse Events (nonserious) regardless of causality is located in the 'Reported Adverse Events' Section.
Time Frame: Up to End of Study (up to approximately Week 39)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | ATYR1940
Number analyzed (Participants) | 8
Participants | 0

8. Primary Outcome: Change From Baseline in Manual Muscle Testing (MMT) Score at Week 12
Description: MMT (muscle strength) will be graded using a modified Medical Research Council scale. Scores were converted to 13-point scale (range from 0 [on contraction palpable] to 12 [normal strength]). An overall total score was calculated by summing all scores for a total possible score of 336. Decreased muscle strength was indicated by a decreased score. An overall total score was calculated as long as 24 of the 28 individual scores were non-missing.
Time Frame: Baseline, Week 12
Population: Cumulative Safety population included all participants who received at least 1 full or partial dose of ATYR1940 in the current study (Study ATYR1940-C-006) and had a post-infusion safety observation since enrollment in parent studies, but with cumulative data from both the parent studies and the current study. Here, 'Number of Participants analyzed' signifies those who were evaluable for this outcome measure and number analyzed signifies those who were evaluable at specified time points only.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ATYR1940
Number analyzed (Participants) | 7
score on a scale
  Baseline | 229.1 (82.56)
  Change at Week 12: number analyzed (Participants) | 6
  Change at Week 12 | 4.3 (13.50)

9. Secondary Outcome: Change From Baseline in Creatinine Kinase at Week 12
Time Frame: Baseline, Week 12
Population: Cumulative Safety population included all participants who received at least 1 full or partial dose of ATYR1940 in the current study (Study ATYR1940-C-006) and had a post-infusion safety observation since enrollment in parent studies, but with cumulative data from both the parent studies and the current study. Here, 'Number of Participants analyzed' signifies those who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units/liter
Arm/Group | ATYR1940
Number analyzed (Participants) | 7
Units/liter | -82.3 (164.98)

ADVERSE EVENTS:
Time Frame: Baseline up to approximately Week 39
Description: Safety population was defined as all participants who received at least 1 full or partial dose of ATYR1940 in the current study (Study ATYR1940-C-006) and had a post-infusion safety observation since enrollment in parent studies. Mortality, Serious Adverse Event, and Other Adverse Event data were prespecified to be collected as a single Arm/Group for any participant who received at least 1 dose of the study drug, regardless of their dose level.
Arm/Group | ATYR1940
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 7/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | ATYR1940 (N=8)
Back pain (Musculoskeletal and connective tissue disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1
Nausea (Gastrointestinal disorders) | 4
Diarrhoea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 2
Cyst (General disorders) | 1
Infusion site pain (General disorders) | 1
Oedema peripheral (General disorders) | 1
Fall (Injury, poisoning and procedural complications) | 4
Back injury (Injury, poisoning and procedural complications) | 1
Bone contusion (Injury, poisoning and procedural complications) | 1
Influenza (Infections and infestations) | 1
Laryngitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Blood bicarbonate decreased (Investigations) | 1
ECG signs of ventricular hypertrophy (Investigations) | 1
Electrocardiogram P wave biphasic (Investigations) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Headache (Nervous system disorders) | 2
Burning sensation (Nervous system disorders) | 1
Tension headache (Nervous system disorders) | 1
Atrioventricular block first degree (Cardiac disorders) | 1
Right atrial dilatation (Cardiac disorders) | 1
Insomnia (Psychiatric disorders) | 1
Ovarian cyst (Reproductive system and breast disorders) | 1/1 — This AE is gender specific.
Rash (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-03-22): https://cdn.clinicaltrials.gov/large-docs/18/NCT02836418/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-19): https://cdn.clinicaltrials.gov/large-docs/18/NCT02836418/SAP_001.pdf